CLINICAL TRIAL: NCT01280643
Title: An Exploratory Study of Chemotherapy for Metastatic Colorectal Cancer Based Upon Thymidine Phosphorylase Expression, KRAS and BRAF Mutation Status, and ERCC1 Expression
Brief Title: Combination Chemotherapy and Cetuximab or Bevacizumab in Treating Patients With Metastatic Colorectal Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB 09-033; NCI-2011-00046 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-01-20; First posted 2011-01-21 (Estimated); Results first posted 2021-03-15 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-02

CONDITIONS: Metastatic Colorectal Cancer
Keywords: stage IVA colon cancer; stage IVA rectal cancer; stage IVB colon cancer; stage IVB rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Fluorouracil; Leucovorin; Oxaliplatin; Irinotecan; Bevacizumab; Cetuximab; Capecitabine; Gene Expression Profiling; Immunohistochemistry; Base Sequence; Polymerase Chain Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- Arm A (Experimental): Patients receive FOLFIRI (FOLolinic acid (leucovorin) Fluorouracil (5-FU) IRInotecan (irinotecan)) chemotherapy comprising fluorouracil intravenously (IV) over 46 hours continuously, leucovorin calcium IV over 2 hours, and irinotecan hydrochloride IV over 90 minutes on days 1 and 15. Patients also receive cetuximab IV over 60-120 minutes on days 1 and 8.
  Interventions: Drug: fluorouracil; Drug: leucovorin calcium; Drug: irinotecan hydrochloride; Biological: cetuximab; Genetic: mutation analysis; Genetic: gene expression analysis; Other: laboratory biomarker analysis; Other: immunohistochemistry staining method; Genetic: nucleic acid sequencing; Genetic: protein expression analysis; Genetic: polymerase chain reaction; Genetic: DNA analysis
- Arm B (Experimental): Patients receive FOLFOX (FOL- Folinic acid (leucovorin) F - Fluorouracil (5-FU) OX - Oxaliplatin (Eloxatin)) chemotherapy comprising fluorouracil IV over 46 hours continuously on day 1 and leucovorin calcium IV over 2 hours and oxaliplatin IV over 2 hours on days 1 and 15. Patients also receive cetuximab IV over 60-120 minutes on days 1 and 8.
  Interventions: Drug: fluorouracil; Drug: leucovorin calcium; Drug: oxaliplatin; Biological: cetuximab; Genetic: mutation analysis; Genetic: gene expression analysis; Other: laboratory biomarker analysis; Other: immunohistochemistry staining method; Genetic: nucleic acid sequencing; Genetic: protein expression analysis; Genetic: polymerase chain reaction; Genetic: DNA analysis
- Arm C (Experimental): Patients receive FOLFIRI chemotherapy as in Arm A and bevacizumab IV over 30-90 minutes on days 1 and 15.
  Interventions: Drug: fluorouracil; Drug: leucovorin calcium; Drug: irinotecan hydrochloride; Biological: bevacizumab; Genetic: mutation analysis; Genetic: gene expression analysis; Other: laboratory biomarker analysis; Other: immunohistochemistry staining method; Genetic: nucleic acid sequencing; Genetic: protein expression analysis; Genetic: polymerase chain reaction; Genetic: DNA analysis
- Arm D (Experimental): Patients receive FOLFOX chemotherapy as in Arm B and bevacizumab IV over 30-90 minutes on days 1 and 15.
  Interventions: Drug: fluorouracil; Drug: leucovorin calcium; Drug: oxaliplatin; Biological: bevacizumab; Genetic: mutation analysis; Genetic: gene expression analysis; Other: laboratory biomarker analysis; Other: immunohistochemistry staining method; Genetic: nucleic acid sequencing; Genetic: protein expression analysis; Genetic: polymerase chain reaction; Genetic: DNA analysis
- Arm E (Experimental): Patients receive CapeIRI (Capecitabine and Irinotecan) chemotherapy comprising capecitabine orally (PO) twice daily (BID) on days 1-14 and irinotecan hydrochloride IV over 90 minutes on days 1 and 8. Patients also receive cetuximab IV over 60-120 minutes on days 1 and 8.
  Interventions: Drug: irinotecan hydrochloride; Biological: cetuximab; Drug: capecitabine; Genetic: mutation analysis; Genetic: gene expression analysis; Other: laboratory biomarker analysis; Other: immunohistochemistry staining method; Genetic: nucleic acid sequencing; Genetic: protein expression analysis; Genetic: polymerase chain reaction; Genetic: DNA analysis
- Arm F (Experimental): Patients receive CapeOX (capecitabine (Xeloda) and oxaliplatin (Eloxatin)) chemotherapy comprising capecitabine PO BID on days 1-14 and oxaliplatin IV over 2 hours on day 1. Patients also receive cetuximab IV over 60-120 minutes on days 1 and 8.
  Interventions: Drug: oxaliplatin; Biological: cetuximab; Drug: capecitabine; Genetic: mutation analysis; Genetic: gene expression analysis; Other: laboratory biomarker analysis; Other: immunohistochemistry staining method; Genetic: nucleic acid sequencing; Genetic: protein expression analysis; Genetic: polymerase chain reaction; Genetic: DNA analysis
- ARM G (Experimental): Patients receive CapeIRI chemotherapy as in Arm E and bevacizumab IV over 30-90 minutes on day 1.
  Interventions: Drug: irinotecan hydrochloride; Biological: bevacizumab; Drug: capecitabine; Genetic: mutation analysis; Genetic: gene expression analysis; Other: laboratory biomarker analysis; Other: immunohistochemistry staining method; Genetic: nucleic acid sequencing; Genetic: protein expression analysis; Genetic: polymerase chain reaction; Genetic: DNA analysis
- Arm H (Experimental): Patients receive CapeOX chemotherapy as in Arm F and bevacizumab IV over 30-90 minutes on day 1.
  Interventions: Drug: oxaliplatin; Biological: bevacizumab; Drug: capecitabine; Genetic: mutation analysis; Genetic: gene expression analysis; Other: laboratory biomarker analysis; Other: immunohistochemistry staining method; Genetic: nucleic acid sequencing; Genetic: protein expression analysis; Genetic: polymerase chain reaction; Genetic: DNA analysis
- Arm I (Experimental): Patients receive treatment as in Arm D.
  Interventions: Drug: fluorouracil; Drug: leucovorin calcium; Drug: oxaliplatin; Biological: bevacizumab; Genetic: mutation analysis; Genetic: gene expression analysis; Other: laboratory biomarker analysis; Other: immunohistochemistry staining method; Genetic: nucleic acid sequencing; Genetic: protein expression analysis; Genetic: polymerase chain reaction; Genetic: DNA analysis

INTERVENTIONS:
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
  Arms: Arm A; Arm B; Arm C; Arm D; Arm I
Drug: leucovorin calcium — Given IV
  Other Names: CF; CFR; LV
  Arms: Arm A; Arm B; Arm C; Arm D; Arm I
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
  Arms: Arm B; Arm D; Arm F; Arm H; Arm I
Drug: irinotecan hydrochloride — Given IV
  Other Names: Campto; Camptosar; CPT-11; irinotecan; U-101440E
  Arms: ARM G; Arm A; Arm C; Arm E
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
  Arms: ARM G; Arm C; Arm D; Arm H; Arm I
Biological: cetuximab — Given IV
  Other Names: C225; C225 monoclonal antibody; IMC-C225; MOAB C225; monoclonal antibody C225
  Arms: Arm A; Arm B; Arm E; Arm F
Drug: capecitabine — Given PO
  Other Names: CAPE; Ro 09-1978/000; Xeloda
  Arms: ARM G; Arm E; Arm F; Arm H
Genetic: mutation analysis — Correlative studies
Genetic: gene expression analysis — Correlative studies
Other: laboratory biomarker analysis — Correlative studies
Other: immunohistochemistry staining method — Correlative studies
  Other Names: immunohistochemistry
Genetic: nucleic acid sequencing — Correlative studies
  Other Names: Gene Sequencing; Molecular Biology, Nucleic Acid Sequencing
Genetic: protein expression analysis — Correlative studies
Genetic: polymerase chain reaction — Correlative studies
  Other Names: PCR
Genetic: DNA analysis — Correlative studies

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fluorouracil, leucovorin calcium, oxaliplatin, capecitabine, and irinotecan hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) and giving the drugs in different combinations may kill more tumor cells. Monoclonal antibodies, such as bevacizumab and cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving combination chemotherapy together with bevacizumab or cetuximab may kill more tumor cells.

PURPOSE:To evaluate the use of standard (KRAS) and experimental (thymidine phosphorylase, ERCC1 and BRAF) tumor testing can aid in selecting chemotherapy regimens

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the feasibility, as defined by completion of three specific marker assays and generation of clinically meaningful endpoints, of selecting treatment regimen components based on biologic tumor characteristics in chemotherapy-naïve patients with metastatic colorectal cancer.

SECONDARY OBJECTIVES:

I. To investigate the response rate associated with genotype/phenotype guided therapy using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

II. To investigate the time to failure of treatment strategy associated with genotype/phenotype guided therapy, defined as the time from initiation of investigational treatment strategy until death, disease progression, initiation of a new therapeutic agent, or disease progression while on a partial or complete treatment holiday.

III. To investigate the progression-free survival associated with genotype/phenotype guided therapy, defined as the time from enrollment to time of progression of disease or death.

OUTLINE: Patients are assigned to treatment groups based on marker assay results.

ARM A: TP-/uncertain, KRAS and BRAF wild-type, ERCC1 high ARM B: TP-/uncertain, KRAS and BRAF wild-type, ERCC1 low/uncertain ARM C: TP-/uncertain, KRAS or BRAF mutant/uncertain, ERCC1 high ARM D: TP-/uncertain, KRAS or BRAF mutant/uncertain, ERCC1 low/uncertain ARM E: TP+, KRAS and BRAF wild-type, ERCC1 high ARM F: TP+, KRAS and BRAF wild-type, ERCC1 low/uncertain ARM G: TP+, KRAS or BRAF mutant/uncertain, ERCC1 high ARM H: TP+, KRAS or BRAF mutant/uncertain, ERCC1 low/uncertain ARM I: TP uninterpretable, KRAS or BRAF uninterpretable, ERCC1 uninterpretable

KRAS testing is standard of care in patients with metastatic colorectal cancer; tymidine phosphorylase, ERCC1 and BRAF testing assays are still experimental.

Courses in arms A-D and arm I repeat every 28 days and courses in arms E-H repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed colon or rectal cancer that has metastasized; no biopsy of metastatic site(s) are required if presentation is consistent with metastatic disease
* Available archived tissue block or slides from the primary colon or rectal cancer; approximately 25 slides from the primary tumor tissue are necessary for testing of all markers
* Patients must have measurable disease by RECIST 1.1, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 10 mm with computed tomography (CT) scan or clinical exam with calipers; lymph nodes must be 15 mm in shortest dimension as measured on CT scan
* Patients may not have received prior therapy for metastatic colorectal cancer; prior adjuvant therapy (including any of the study agents) is permitted if completed > 6 months from the initial detection of metastatic disease
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 2 X institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/ alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) =< 3 X institutional ULN or =< 5 X ULN if known liver metastases
* Creatinine clearance >= 50 mL/min (as calculated by Cockroft and Gault formula)
* Urine protein:creatinine (UPC) ratio < 1.0 at screening (as calculated from urine protein concentration and urine creatinine concentration); patients with a UPC ratio >= 1 will undergo a 24-hour urine collection, which must be adequate and demonstrate < 1 gram in order to participate
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had previous chemotherapy for metastatic colorectal cancer
* Uncontrolled hypertension (>150/100 mmHg) despite a stable regimen of anti-hypertensive medication
* History of cardiovascular disease, defined as previous myocardial infarction, cerebrovascular accident, uncontrolled congestive heart failure (New York Heart Association > Class II), clinically significant ventricular arrhythmia requiring medication, clinically significant peripheral vascular disease, or unstable angina within 6 months of study enrollment
* Underlying neuropathy >= grade 2
* Serious non-healing wounds, ulcers, or fistulas
* Major surgery, open biopsy, or major traumatic injury within 28 days of registration, or anticipation of need for surgical procedure during course of study, and core biopsy or fine needle aspiration within 7 days of registration; closed biopsy or access port placement is acceptable
* A history of thrombotic or hemorrhagic disorder; patients with elevated international normalized ratio (INR) (2.0 to 3.0) on stable doses of therapeutic anticoagulation are eligible
* Untreated brain metastases; patients with treated brain metastases who have completed radiation therapy, are clinically and radiographically stable, and are off steroid therapy may be enrolled
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cetuximab, oxaliplatin, capecitabine, or other agents used in the study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded; breastfeeding should be discontinued if the mother is treated with chemotherapy
* Human Immunodeficiency Virus (HIV)-positive patients on combination antiretroviral therapy are ineligible; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Patients must not have a history of another neoplasm < 5 years prior to enrollment, except for non-metastatic, non-melanoma skin cancer or carcinoma in situ of the cervix
* Patients of child-bearing potential who are unwilling or unable to utilize contraceptive measures including barrier contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Crystal Denlinger, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F | ARM G | Arm H | Arm I
Started | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study closed prematurely due to poor accrual
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F | ARM G | Arm H | Arm I | Total
Number analyzed (Participants) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0 | 0 |  |  |  |  |  | 0
  Between 18 and 65 years |  | 1 | 0 | 1 |  |  |  |  |  | 2
  >=65 years |  | 0 | 1 | 0 |  |  |  |  |  | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 0 | 0 | 0 |  |  |  |  |  | 0
  Male |  | 1 | 1 | 1 |  |  |  |  |  | 3
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1 | 1 |  |  |  |  |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Feasibility, Defined as a Sufficient Proportion of Subjects Having Available Tissue and an Acceptable Composite Assay Success Rate Among Tested Subjects
Time Frame: Over 21 months
Population: Too few enrolled participants for meaningful analysis
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F | ARM G | Arm H | Arm I
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Best Overall Response Via RECIST
Time Frame: Over 21 months
Population: Too few enrolled participants for meaningful analysis
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F | ARM G | Arm H | Arm I
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Time to Failure of Treatment Strategy
Time Frame: Over 21 months
Population: Too few enrolled participants for meaningful analysis
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F | ARM G | Arm H | Arm I
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Progression-free Survival
Time Frame: Over 21 months
Population: Too few enrolled participants for meaningful analysis
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F | ARM G | Arm H | Arm I
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: No patients accrued to arms A, E, F, G, H, I due to premature study closure resulting from slow accrual
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F | ARM G | Arm H | Arm I
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1 | 1/1 | 0/1 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 1/1 | 0/1 | 0/1 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 1/1 | 1/1 | 1/1 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=0) | Arm B (N=1) | Arm C (N=1) | Arm D (N=1) | Arm E (N=0) | Arm F (N=0) | ARM G (N=0) | Arm H (N=0) | Arm I (N=0)
Hospitalization - Chest pain (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=0) | Arm B (N=1) | Arm C (N=1) | Arm D (N=1) | Arm E (N=0) | Arm F (N=0) | ARM G (N=0) | Arm H (N=0) | Arm I (N=0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | NA | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea/Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysguesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sour stomach (General disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Bilateral hands
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parasthesias (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — In hands and feet
Pain (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restless legs (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Cramping in legs
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushed face (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Jaw pain
Pharyngitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Scratchy throat
Insomnia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Twitching/restlessness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — At injection site
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Too few enrolled participants for meaningful analysis. Study closed prematurely due to slow accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No